CLINICAL TRIAL: NCT04272502
Title: Phase I Clinical Trial to Compare the Pharmacokinetics and Safety of CKD-348 in Healthy Adult Volunteers
Brief Title: Clinical Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-348 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A86_02BE1902P
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence A (Experimental): CKD-828, D326, D337, CKD-F1, CKD-F2
  Interventions: Drug: CKD-348 F1, CKD-348 F2, CKD-828, D326, D337
- Sequence B (Experimental): CKD-828, D326, D337, CKD-F1, CKD-F2
  Interventions: Drug: CKD-348 F1, CKD-348 F2, CKD-828, D326, D337
- Sequence C (Experimental): CKD-828, D326, D337, CKD-F1, CKD-F2
  Interventions: Drug: CKD-348 F1, CKD-348 F2, CKD-828, D326, D337

INTERVENTIONS:
Drug: CKD-348 F1, CKD-348 F2, CKD-828, D326, D337 — Each arm has a different order for taking IP

SUMMARY:
Phase I clinical trial to compare the pharmacokinetics and safety of CKD-348 with co-administration of CKD-828, D326 and D337 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. 19 ≤ age ≤ 45
2. Health Volunteers
3. Subject who agreeds to participate in this clinical trial voluntarily

Exclusion Criteria:

1. Subject who cannot participate in a clinical trial based on the PI's judgment

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 hour ~ 144 hour
  Maximum plasma concentration of the drug
AUCt | 0 hour ~ 144 hour
  Area under the concentration-time curve from time zero to time

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No